CLINICAL TRIAL: NCT06304948
Title: The Link Between Human Cytomegalovirus Gene Expression and Glutamate Levels in Migraine :Relationship to the Vit D Deficiency
Brief Title: The Link Between Human Cytomegalovirus Gene Expression and Glutamate Level in Migraine;Relation to Vitamin D Deficiency
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Omar Ali, Doctor resident, Assiut University
Other Study IDs: Vitamin D and migraine
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To correlate serum 25(OH)-vitamin D level with duration, frequency, and severity of migraine headache attacks
2. To evaluate the relationship between the serum level of vitamin D and other indices in patients with migraine.
3. To correlate the serum level of glutamate with gene expression of in migraine

DETAILED DESCRIPTION:
According to the report of global burden of disease (GBD) 2016, migraine headache has been established as the leading disability cause in the globe among under 50 years old [1]. It has been estimated that migraine affects about 11% of adults with a major impact on those aged between 25 to 55 years, which consequently lead to the high headache burden on individuals, communities, health care systems, and societies. Migraine is 2-3 times more common in women than in men. Migraine attacks are usually more prolonged, with higher intensity and more disability among females.

Current pharmacological treatments for migraine demonstrated limited efficacy in some patients and commonly lead to some adverse events such as weight reduction or weight gain, fatigue/sleepiness, sweating, night dreams, gastrointestinal upset and hypotension or reduced concentration. Novel therapeutic approaches of nutritional agents have become the promising strategies to alleviate symptoms of migraine. Vitamin D, one of the dietary agents, has revealed some potential in managing pain and migraine.

Cytomegalovirus (CMV) contamination is one of the clinically most critical irresistible complications of solid-organ transplantation. CMV disease, characterized as a critical rise within the titer of CMV-specific antibodies, happens in 44 % to 85% of kidney, heart, and liver transplant recipients - basically within the to begin with 3 months post transplantation, when immunosuppression is most intense. CMV malady shows in transplant beneficiaries essentially within the organ transplanted with the chance of successive dispersal and disability of other organs such as the central-nervous system, eye, and urogenital- or gastrointestinal tract. Additionally, dynamic CMV disease could be a noteworthy autonomous indicator of intense unite dismissal and event of artful contaminations.

Join brokenness and dismissal are related with vitamin D (VD) lack. In patients with end-stage organ disappointment anticipating transplant, VD lacking and lack are greatly common. Inadequately levels of vitamin D metabolites (25-hydroxyvitamin D [25(OH)D3] and 1,25-hydroxyvitamin D [1a,25_ Dihydroxyvitamin D3] have been detailed for patients with terminal congestive heart disappointment. pneumonic infection, liver disappointment [5], and incessant kidney illness.

in the past few years, there has been increasing interest in the complex interplay between vitamin D and infectious pathogens 7 Vitamin D supplementation is beneficial for patients with HIV, hepatitis C virus, Chlamydia spp. or mycobacterial infection. A significant reduction in the risk of CMV infection and disease by vitamin D supplementation would be highly attractive because of a high therapeutic index of vitamin D, the ease of application (oral solutions), and added benefits such as improved musculoskeletal health. Contrary to expectation, we found that CMV infection interferes with the vitamin D system of mammalian cells.

CMV infection downregulated vitamin D receptor expression and this downregulation was specific for CMV and was not observed for other, common human viruses. This observation may have far-reaching virological, immunological, and clinical implication

The aim of the present study was to assess a possible effect of migraine in patients with CMV infection on vit D levels and Glutamate levels to combine existing knowledge about the role of glutamate in migraine pathogenesis along with information on nutrients that are protective against glutamate excitotoxicity, and then end with a proposed dietary treatment for migraine management.

There is an obvious gap between our understanding of migraines and the dietary strategies which have been administered so far, since dietary nutrients are often studied separately, and no specific diet for migraine has been developed. However, the beneficial effects of the low glutamate diet on widespread chronic pain disorders appear to have overlapping mechanistic effects, and additionally is some preliminary evidence supporting an effect on migraine. Thus, further research on this dietary strategy in migraine is warranted

ELIGIBILITY:
Inclusion Criteria:

1. Selected patients fulfilled the criteria for diagnosis of migraine headache based on International Classification of Headache Disorders-II (ICHD-II) diagnostic criteria.
2. The age of the selected patients ranged between 15 and 55 years of both sexes
3. Able to give informed consent.

Exclusion Criteria:

* b. Exclusion criteria:

  1. presence of neurological disease other than migraine
  2. presence of other chronic medical conditions
  3. Participants in both groups were excluded from the study if they consumed vitamin D supplements in the preceding 3 months (any dose); or if they were taking medications that could affect vitamin D serum level such as glucocorticoids, thiazide diuretics, or statins. 4)patients refuse to participate in the study

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Selected patients fulfilled the criteria for diagnosis of migraine headache based on International Classification of Headache Disorders-II (ICHD-II) diagnostic criteria.
  And The age of the selected patients ranged between 15 and 55 years of both sexes
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
The Link between human cytomegalovirus gene expression and glutamate levels in Migraine :relationship to the Vit D Deficiency | Baseline
  Relation between CMV infection and glutamate level in patients with migraine in relation to vitamin D level

CONTACTS AND LOCATIONS:
Overall Officials: Essam S Darweish, Study Director — Assuit u

REFERENCES:
- [Background] Steiner TJ, Stovner LJ, Vos T, Jensen R, Katsarava Z. Migraine is first cause of disability in under 50s: will health politicians now take notice? J Headache Pain. 2018 Feb 21;19(1):17. doi: 10.1186/s10194-018-0846-2. No abstract available. PMID 29468450
- [Background] Steininger C. Clinical relevance of cytomegalovirus infection in patients with disorders of the immune system. Clin Microbiol Infect. 2007 Oct;13(10):953-63. doi: 10.1111/j.1469-0691.2007.01781.x. PMID 17803749
- [Background] Hartmann A, Sagedal S, Hjelmesaeth J. The natural course of cytomegalovirus infection and disease in renal transplant recipients. Transplantation. 2006 Jul 27;82(2 Suppl):S15-7. doi: 10.1097/01.tp.0000230460.42558.b0. PMID 16858268
- [Background] Monegal A, Navasa M, Guanabens N, Peris P, Pons F, Martinez de Osaba MJ, Rimola A, Rodes J, Munoz-Gomez J. Bone mass and mineral metabolism in liver transplant patients treated with FK506 or cyclosporine A. Calcif Tissue Int. 2001 Feb;68(2):83-6. doi: 10.1007/BF02678145. PMID 11310351
- [Background] Latic N, Erben RG. Vitamin D and Cardiovascular Disease, with Emphasis on Hypertension, Atherosclerosis, and Heart Failure. Int J Mol Sci. 2020 Sep 4;21(18):6483. doi: 10.3390/ijms21186483. PMID 32899880
- [Background] Gallo D, Mortara L, Gariboldi MB, Cattaneo SAM, Rosetti S, Gentile L, Noonan DM, Premoli P, Cusini C, Tanda ML, Bartalena L, Piantanida E. Immunomodulatory effect of vitamin D and its potential role in the prevention and treatment of thyroid autoimmunity: a narrative review. J Endocrinol Invest. 2020 Apr;43(4):413-429. doi: 10.1007/s40618-019-01123-5. Epub 2019 Oct 4. PMID 31584143
- [Background] Kearns MD, Alvarez JA, Seidel N, Tangpricha V. Impact of vitamin D on infectious disease. Am J Med Sci. 2015 Mar;349(3):245-62. doi: 10.1097/MAJ.0000000000000360. PMID 25334038
- [Background] Wells RE, Beuthin J, Granetzke L. Complementary and Integrative Medicine for Episodic Migraine: an Update of Evidence from the Last 3 Years. Curr Pain Headache Rep. 2019 Feb 21;23(2):10. doi: 10.1007/s11916-019-0750-8. PMID 30790138
- [Background] Gazerani P, Fuglsang R, Pedersen JG, Sorensen J, Kjeldsen JL, Yassin H, Nedergaard BS. A randomized, double-blinded, placebo-controlled, parallel trial of vitamin D3 supplementation in adult patients with migraine. Curr Med Res Opin. 2019 Apr;35(4):715-723. doi: 10.1080/03007995.2018.1519503. Epub 2018 Sep 28. PMID 30182753